CLINICAL TRIAL: NCT02060370
Title: A Phase II Study of Alternative Sunitinib Scheduling in Patients With Metastatic Renal Cell Carcinoma (mRCC)
Brief Title: Sunitinib Scheduling in Metastatic Renal Cell Carcinoma (mRCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0944; NCI-2014-01908 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-02-10; First posted 2014-02-12 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Genitourinary Cancer; Kidney Cancer
Keywords: Genitourinary Cancer; Kidney Cancer; Metastatic Renal Cell Carcinoma; mRCC; Sunitinib; Sunitinib malate; SUO11248; Sutent; Questionnaire; Survey
MeSH Terms: conditions — Urogenital Neoplasms; Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Sunitinib; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sunitinib (Experimental): Sunitinib starting dose 50 mg by mouth daily given for 2 weeks "on" followed by 1 week "off". 1 cycle is 6 weeks.
  Interventions: Drug: Sunitinib; Behavioral: Questionnaire

INTERVENTIONS:
Drug: Sunitinib — Starting dose: 50 mg by mouth daily given for 2 weeks "on" followed by 1 week "off". 1 cycle is 6 weeks.
  Other Names: Sunitinib Malate; SUO11248; Sutent
Behavioral: Questionnaire — Questionnaire completion on Day 1 of Cycle 1, and on Day 35 of Cycles 2, 4, and 6.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is to learn more about the safety of giving sunitinib to patients with metastatic kidney cancer for 2 weeks followed by 1 week in which they receive no drug. Researchers want to learn more about the side effects of the drug and the effects of a different dosing schedule.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will take sunitinib capsules by mouth every day for 2 weeks, followed by 1 week in which you do not receive any study drug. This will then be repeated every 3 weeks.

Every 6 weeks will be 1 study cycle.

If you have any side effects tell the study doctor right away. The study doctor may change your dose of the study drug.

Study Visits:

Every day during the first week, and then at least 1 time each week during the study, your blood pressure will be checked (either at home, at the clinic, or by your local doctor). You will need to write down your blood pressure in a blood pressure diary each time you check it and bring the diary with you to each clinic visit.

On Day 1 of Cycle 1:

* You will have a physical exam.
* Blood (about 3-4 tablespoons) will be drawn for routine and biomarker testing.
* You will fill out a questionnaire about the quality of your life and about how you are feeling. This should take about 5 minutes.

On Day 42 of every cycle:

* You will have a physical exam.
* Blood (about 3-4 tablespoons) will be drawn for routine tests.

On Day 42 of every even-numbered cycle (Cycles 2, 4, 6, and so on):

* You will have a CT scan of your chest, abdomen, and pelvis.
* Blood (about 1 tablespoon) will be drawn to check your thyroid function.
* Blood (about 2 tablespoons) will be drawn for biomarker testing. (Cycles 2 , 4, and 6 only)
* You will fill out the questionnaire about the quality of your life and about how you are feeling. (Cycles 2 , 4, and 6 only)

At any time that the doctor thinks it is needed, additional blood (about 1 tablespoon) may be drawn to check your thyroid function, and you may need to have a bone scan and CT scan or MRI of the brain to check the status of the disease.

Length of Study:

You may continue taking the study drug for as long as the study doctor thinks it is in your best interest. You will be taken off treatment if the disease gets worse, intolerable side effects occur, or if you are unable to follow study directions.

Your participation in this study will be over after the follow-up visit. However, the study team may perform a medical record review or follow-up call to check on how you are doing. If you are called, this should last about 5-10 minutes.

End-of-Treatment Visit:

After you are no longer receiving the study drug, you will have an end-of-treatment visit. You will have a physical exam and blood (about 3-4 tablespoons) will be drawn for routine and biomarker testing.

End-of- Treatment Follow-Up Visit:

About 30 days after your end-of-treatment visit you will have a follow-up visit and the following procedures will be performed:

* You will have a physical exam.
* Blood (about 3-4 tablespoons) will be drawn for routine tests.
* You will have CT scans of your chest, abdomen and pelvis to check the status of the disease.

This is an investigational study. Sunitinib is FDA approved and commercially available to treat advanced kidney cancer. The dosing schedule being used on this study is investigational.

Up to 60 participants will be enrolled in this study. Up to 60 may take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically-confirmed metastatic renal cell carcinoma of clear cell histology. Prior nephrectomy is not a requirement for eligibility
2. Age >/=18 years
3. Measurable or evaluable metastatic disease per RECIST v 1
4. ECOG performance status 0-1
5. Normal organ and bone marrow function as defined by: Serum aspartate transaminase (AST) or serum glutamic oxaloacetic transaminase (SGOT) and serum alanine transaminase (ALT) or serum glutamic pyruvic transaminase (SGPT) </= 2.5 x laboratory upper limit of normal (ULN); Total serum bilirubin </= 2.0 x ULN; Absolute neutrophil count (ANC) >/= 1500/µL; Platelets >/= 100,000/µL; Hemoglobin >/= 9.0 g/dL (transfusion permitted); Serum calcium </= 12.0 mg/dL; Serum creatinine </= 2.5 mg/dL
6. Patients with a history of deep venous thromboembolism or pulmonary embolism on treatment with anticoagulation are eligible for the study.
7. Subjects must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Prior treatment with sunitinib or any other systemic therapy in the metastatic setting (prior neo/adjuvant therapy will be allowed if completed > 6 months prior to registration and therapy not discontinued for toxicity)
2. Uncontrolled hypertension (defined as blood pressure >140/90 mm Hg not controlled with anti-hypertensives)
3. Prior intraabdominal, intrathoracic, vascular, spinal or intracranial surgery or radiation therapy within 4 weeks of starting treatment
4. History of or known brain metastases, spinal cord compression, or carcinomatous meningitis
5. New York Heart Association (NYHA) grade II or greater congestive heart failure
6. Current treatment on another therapeutic clinical trial
7. Any of the following within the preceding 6 months- myocardial infarction, severe/unstable angina, severe peripheral vascular disease (claudication) or procedure on peripheral vasculature, coronary/peripheral artery bypass, graft, cerebrovascular accident or transient ischemic attack, clinically significant bleeding
8. Pregnant or breastfeeding women are excluded from this study because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with sunitinib. Breastfeeding must be discontinued if the mother is treated with sunitinib
9. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness
10. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with sunitinib. In addition, these patients are at increased risk of lethal infections when treated with marrow suppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jonasch, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - Stanford University Medical Center, Stanford, California
  - Lineberger Cancer Center, Chapel Hill, North Carolina
  - Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Jonasch E, Slack RS, Geynisman DM, Hasanov E, Milowsky MI, Rathmell WK, Stovall S, Juarez D, Gilchrist TR, Pruitt L, Ornstein MC, Plimack ER, Tannir NM, Rini BI. Phase II Study of Two Weeks on, One Week off Sunitinib Scheduling in Patients With Metastatic Renal Cell Carcinoma. J Clin Oncol. 2018 Jun 1;36(16):1588-1593. doi: 10.1200/JCO.2017.77.1485. Epub 2018 Apr 11. PMID 29641297
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty participants enrolled between August 2014 and March 2016. Participants recruited from The University of Texas MD Anderson Cancer Center, Cleveland Clinic Foundation, Fox Chase Cancer Center, and University of North Carolina Lineberger Cancer Center). All participants had confirmed treatment naive metastatic clear cell renal cell carcinoma.
Pre-assignment Details: One participant did not take the study medication due to declining mental health status before the first dose was initiated. Consequently, only 59 patients were included in the final analysis.
Groups:
- Alternating Sunitinib: Starting dose of 50 mg by mouth daily for 2 weeks followed by 1 week of no drug. 1 cycle equaled six weeks.
Period: Overall Study
Arm/Group | Alternating Sunitinib
Started | 60
Completed | 59
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 65 [45 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 50
  More than one race | 0
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  United States | 60
Memorial Sloan Kettering Cancer Center (MSKCC) Risk Factor [Count of Participants; unit: Participants] — Method used to predict survivability of participants at outset of treatment
  Participants
    Good | 13
    Intermediate | 40
    Poor | 6
    Unknown | 1
Number of Metastatic Sites [Median (Full Range); unit: Number of metastatic sites] — Describes the extent of the participants' advance disease
  Number of metastatic sites | 2 [1 to 4]
Metastatic Sites [Count of Participants; unit: Participants]
  Lung | 39
  Lymph node | 10
  Liver | 8
  Bone | 3
  Other | 29

OUTCOME MEASURES:

1. Primary Outcome: Rate of Toxicity
Description: Determine the number of participants who experience a specific, treatment-related adverse events at a grade three, four or five: fatigue, hand-foot syndrome, and/or diarrhea. Adverse events as defined by the Common Terminology Criteria for Adverse Events (CTCAE) version 4
Time Frame: Participants were monitored for toxicities for 30 days after treatment was discontinued; total treatment duration approximately 34 months
Measure: Count of Participants; unit: Participants
Arm/Group | Alternating Sunitinib
Number analyzed (Participants) | 59
Participants
  Grade>=3, of all 3 adverse events | 15
  Fatigue, Grade >=3 | 8
  Diarrhea, Grade >=3 | 5
  Hand-foot syndrome, Grade >=3 | 3

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 17 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alternating Sunitinib
Number analyzed (Participants) | 59
months | 13.7 [10.9 to 16.3]

3. Secondary Outcome: The Number and Percentage of Participants Who Experienced a Grade 3, 4, or 5 Adverse Event
Description: Adverse events as defined by Common Terminology Criteria for Adverse Events (CTCAE) version 4
Time Frame: Participants were monitored for toxicities for 30 days after treatment was discontinued or until death, whichever occurred first.
Measure: Count of Participants; unit: Participants
Arm/Group | Alternating Sunitinib
Number analyzed (Participants) | 59
Participants
  Any grade ≥3 event | 35
  Alkaline phosphatase increased | 1
  Anemia | 6
  Dehydration | 1
  Diarrhea | 5
  Fatigue | 8
  Pancreatic insufficiency | 1
  Headache | 1
  Hypertension | 16
  Hyponatremia | 2
  Hypophosphatemia | 1
  Lymphocyte count decreased | 1
  Mucositis oral | 5
  Gout | 1
  Neutrophil count decreased | 8
  Hand-foot syndrome | 3
  Platelet count decreased | 2
  Thromboembolic event | 3
  Urticaria | 1
  Vascular access complication | 1
  Vomiting | 1
  White blood cell decreased | 4

4. Secondary Outcome: Dose Reductions and Treatment Discontinuations Due to Unacceptable Toxicities
Description: Reported as the number and percentage of participants who underwent one or more dose reductions, as well as, the number and percentage of participants whose treatment ended.
Time Frame: 2 years
Population: Out of the 59 participants only 29 encountered a dose reduction. The number of dose reductions a participant experienced was also reported with the percentage being based on the 29 participants who had a reduction.
Measure: Count of Participants; unit: Participants
Arm/Group | Alternating Sunitinib
Number analyzed (Participants) | 59
Participants
  1 Dose Reduction | 7
  2 Dose Reductions | 14
  3 Dose Reductions | 3
  4 Dose Reductions | 5

5. Secondary Outcome: Changes in Participant Reported Outcomes in the Functional Assessment of Cancer Therapy-General (FACT-G)
Description: Participants completed FACT-G suveys evaluating quality of life at weeks 0, 12, 24, and 36. The score range is from 0 to 180 with higher scores reflecting a better quality of life. The results were reported for each time point for all participants and then broken into two groups: participants with a grade 3 toxicity and participants without a grade 3 toxicity. The total number of surveys changes as the weeks progress.
Time Frame: 36 weeks from the start of treatment
Population: The number of surveys collected at week 0, 12,24, and 36 are 54, 49, 44, and 35 surveys.The number of surveys with a grade 3 toxicity collected at week 0, 12, 24, and 36 are 14, 11, 12, and 10 surveys. The number of surveys without a grade 3 toxicity collected at week 0, 12, 24, and 36 are 40, 38, 32, and 25 surveys.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Alternating Sunitinib
Number analyzed (Participants) | 54
Score on a scale
  All Participants- week 0 | 87.8 [57.7 to 108]
  All Participants- week 12 | 88 [46 to 106]
  All Participants- week 24 | 86 [44 to 108]
  All Participants- week 36 | 89 [61 to 106]
  Grade 3 tox - week 0 | 86.8 [56 to 108]
  Grade 3 tox - week 12 | 79.5 [46 to 100]
  Grade 3 tox - week 24 | 79 [44 to 106]
  Grade 3 tox - week 36 | 83 [63 to 106]
  No grade 3 tox - week 0 | 88.8 [52.7 to 105]
  No grade 3 tox - week 12 | 89.8 [46.8 to 106]
  No grade 3 tox - week 24 | 91.8 [55.2 to 108]
  No grade 3 tox - week 36 | 93.8 [61 to 104]

6. Secondary Outcome: Changes in Circulating DNA Levels With Antiangiogenic Treatment
Time Frame: Not applicable due data not generated due to timing and budgetary issues
Population: Data were not collected due to timing and budgetary issues.
Arm/Group | Alternating Sunitinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Toxicities were monitored from the first dose until 30 days after the last dose of study drug was given, monitoring was approximately 36 months.
Arm/Group | Sunitinib
All-Cause Mortality (participants affected / at risk) | 2/59
Serious Adverse Events (participants affected / at risk) | 35/59
Other Adverse Events (participants affected / at risk) | 59/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=59)
Alkaline phosphatase increased (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 8
Diarrhea (Gastrointestinal disorders) | 5
Pancreatic insufficiency (Endocrine disorders) | 1
Headache (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 16
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1
Lymphocyte count decreased (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 5
Gout (Metabolism and nutrition disorders) | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 8
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 3
Platelet count decreased (Blood and lymphatic system disorders) | 2
Thromboembolic event (Vascular disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1
Vascular access complication (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
White blood cell decreased (Blood and lymphatic system disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=59)
Abdominal pain (Gastrointestinal disorders) | 3
Alanine aminotransferase increased (Investigations) | 11
Alkaline phosphatase increased (Investigations) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 3
Anal mucositis (Gastrointestinal disorders) | 4
Anemia (Blood and lymphatic system disorders) | 32
Anorexia (Gastrointestinal disorders) | 12
Aspartate aminotransferase increased (Investigations) | 19
Bloating (Gastrointestinal disorders) | 3
Blood bilirubin increased (Investigations) | 6
CD4 lymphocytes decreased (Investigations) | 3
Constipation (Gastrointestinal disorders) | 6
Creatinine increased (Investigations) | 21
Diarrhea (Gastrointestinal disorders) | 45
Dry mouth (Gastrointestinal disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 4
Dysesthesia (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 27
Dyspepsia (Gastrointestinal disorders) | 13
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12
Edema (General disorders) | 9
TSH increased (Endocrine disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Fatigue (General disorders) | 49
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7
Headache (Nervous system disorders) | 6
Hemoglobinuria (Renal and urinary disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypertension (Vascular disorders) | 10
Hypoalbuminemia (Metabolism and nutrition disorders) | 12
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 5
Hypothyroidism (Endocrine disorders) | 15
Lymphocyte count decreased (Blood and lymphatic system disorders) | 7
Mucositis oral (Gastrointestinal disorders) | 32
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Nausea (Gastrointestinal disorders) | 26
Neutrophil count decreased (Blood and lymphatic system disorders) | 23
Non-cardiac chest pain (General disorders) | 4
Oral dysesthesia (Gastrointestinal disorders) | 8
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 32
Rash (Skin and subcutaneous tissue disorders) | 24
Paresthesia (Nervous system disorders) | 4
Platelet count decreased (Investigations) | 36
Proteinuria (Renal and urinary disorders) | 23
Pruritus (Skin and subcutaneous tissue disorders) | 8
Hair hypopigmentation (Skin and subcutaneous tissue disorders) | 4
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 12
Thromboembolic event (Vascular disorders) | 3
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 3
Vomiting (Gastrointestinal disorders) | 14
Watering eyes (Eye disorders) | 10
Weight loss (Investigations) | 8
White blood cell decreased (Blood and lymphatic system disorders) | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT02060370/Prot_SAP_000.pdf